CLINICAL TRIAL: NCT04372472
Title: SQuISH-COVID: A Pilot Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Cytovale, Inc. (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: CV-CLN-003
Record Dates: First submitted 2020-04-29; First posted 2020-05-04 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-06

CONDITIONS: Sepsis; COVID-19
Keywords: Sepsis; COVID
MeSH Terms: conditions — Sepsis; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

SUMMARY:
This is a single-site prospective study to evaluate the diagnostic performance of the investigational SeptiScan System for patients presenting to the Emergency Department with signs or suspicion of COVID-19 or other infectious respiratory diseases.

ELIGIBILITY:
Inclusion Criteria:

Subjects meeting the following criteria may be eligible for participation in the study:

1. ≥ 18 years old or older
2. The first vital sign (any one of: blood pressure, temperature, pulse or respiratory rate) has been recorded in the medical record
3. A complete blood count has been ordered for which a blood sample has been collected within 4.5 hours since the first vital sign was recorded
4. Signs or suspicion of a respiratory infection, defined as:

   1. Subject designated for evaluation in the ED respiratory or pulmonary pod or similar location. OR
   2. An order placed for a respiratory viral panel. OR
   3. An order placed for a SARS-CoV-2 test. OR
   4. A subject self-reported as having tested positive for the SARS-CoV-2 test within the previous 7 days and returning with a related complaint.

Exclusion Criteria:

Subjects are excluded from study participation if they meet any of the following criteria:

a. Blood sample volume is < 300 ul; insufficient quantity for SeptiScan testing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enroll up to 300 participants from the emergency department at one clinical research site. Subjects who are suspected of having COVID-19 or other infectious respiratory diseases may be eligible for the study.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2020-04-07 (Actual); Primary Completion 2020-08-14 (Actual); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
To demonstrate the performance of the SeptiScan System as a diagnostic marker of life-threatening organ dysfunction caused by a dysregulated host immune response to infection. | Day of enrollment through Day 5
  The SeptiScan System is an investigational microfluidic assay that measures the biophysical properties of human leukocytes as an aid, in conjunction with other clinical assessments, to detect life-threatening organ dysfunction caused by a dysregulated host immune response to infection. The SeptiScan System score is presented in three Interpretation Bands of low, intermediate, and high probability of disease. Remnant blood samples will be obtained from subjects in Emergency Department with signs or suspicion of COVID-19 or other infectious respiratory diseases. The blood samples will be analyzed using the SeptiScan System.

CONTACTS AND LOCATIONS:
Overall Officials: Hollis R O'Neal, Jr., MD, MSc, Principal Investigator — Pulmonary & Critical Care LSUHSC, Baton Rouge
Locations (1):
- Our Lady of the Lake Regional Medical Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No